CLINICAL TRIAL: NCT02439359
Title: A Phase 1, Placebo-Controlled, Dose-Escalating Study to Examine the Safety and Tolerability of Single Intravenous Doses of CF-301 in Healthy Male and Female Subjects
Brief Title: A Placebo-Controlled, Dose-Escalating Study to Examine the Safety and Tolerability of Single Intravenous Doses of CF-301 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ContraFect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF 301-101
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2016-12

CONDITIONS: Staphylococcus Aureus Bloodstream Infections (BSI; Bacteremia)
MeSH Terms: conditions — Bacteremia | interventions — exebacase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- CF-301 (Experimental): CF-301
  Interventions: Drug: CF-301

INTERVENTIONS:
Drug: CF-301 — Dose escalation
  Arms: CF-301
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Phase 1, Placebo-Controlled, Dose-Escalating Study to Examine the Safety and Tolerability of Single Intravenous Doses of CF-301 in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy male of any race or ethnicity, at least 18 years of age and no more than 55 years of age, inclusively, OR
2. Be a healthy female of any race or ethnicity of non-childbearing potential between 18 and 55 years of age, inclusive. OR
3. Be a healthy non-pregnant, non-lactating female of any race or ethnicity of childbearing potential between 18 and 55 years of age,
4. Contraception in use for at least 60 days prior to the Screening visit,
5. Have a body mass index (BMI) between 18.5 and 32 kg/m2, inclusive
6. Have no significant diseases in the opinion of the Investigator in the medical history or clinically significant findings on physical examination or clinical laboratory evaluations.

Exclusion Criteria:

1. Any disease or condition in the opinion of the Investigator that might compromise the cardiovascular, hematologic, renal, hepatic, pulmonary (including chronic asthma), endocrine (eg, diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
2. The presence of clinically significant laboratory values that are out of the normal range.

   - Subjects with an aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), alkaline phosphatase, bilirubin, blood urea nitrogen (BUN), creatinine, prothrombin time (PT), or activated partial thromboplastin time (aPTT) > 5% above the upper limit of normal, or hemoglobin or hematocrit level < 5% below the lower limit of normal may not be enrolled.
3. A history of alcoholism or drug addiction, or illicit drug use within the past 2 years, or positive results from a urine screen for substances of abuse.
4. Has smoked within 28 days prior to receiving study drug or has a positive urine test for cotinine.
5. A history of serious mental illness.
6. A history of difficulty donating blood or inadequate venous access.
7. The donation of blood or plasma within 28 days prior to receiving study drug.
8. A positive hepatitis screen that tests for both hepatitis B surface antigen (HBsAg) and antibody to hepatitis C virus (HCVAb).
9. A positive test result for human immunodeficiency virus (HIV) antibody by enzyme immunoassay, which is confirmed by Western blot.
10. Use of an investigational drug or product, or participation in a drug study within a period of 28 days prior to receiving study drug (for investigational drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
11. Use of any prescription or over-the-counter (OTC) drug therapy, including herbal, homeopathic, vitamins, minerals and nutritional supplements, within 2 weeks prior to receiving the study drug contraceptives in women of childbearing potential is allowed during the study.

    - If a subject taking prescription drug therapy for chronic diseases, but that prescription is stopped in order to qualify for the study, the subject should not be enrolled in the study.
12. Use of any drug therapy (ie, prescription drugs, over-the counter products, herbal and vitamin products) known to induce or inhibit cytochrome P450 hepatic enzymes responsible for drug metabolism within 28 days prior to receiving study drug or during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by AE's | up to 8 months
  Safety and tolerability will be assessed by monitoring AEs and performing physical/clinical examinations.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lenexa, Kansas
  - Cf 301-105, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Public Presentation at ECCMID April 2016